CLINICAL TRIAL: NCT05966779
Title: Physical Therapy Intervention in the Immediate Postoperative Phase of Lipedema Surgery
Brief Title: Physical Therapy in Lipedema Surgery
Status: Completed | Type: Observational
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Ester Cerezo-Téllez, PhD., Professor, University of Alcala
Other Study IDs: OE36/2023
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Assessment; Lipedema; Vascular Diseases; Dermatologic Complication
Keywords: Lipedema, physical therapy,liposuction,complications,treatment,assessment
MeSH Terms: conditions — Lipedema; Vascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- modified CDT physical therapy protocol, based on Godoy's Method: A complete physical therapy assessment was done. All sociodemographic data were recruited as well as body mass index (BMI), the month of intervention, kind of surgery, extracted liters, psychological treatment, physical therapy sessions, pain, mobility, complications (seroma, wound infection, chafing or risk of ulcer, pain, fibrosis, genital edema), compression, smoking, satisfaction with the treatment received.
  A modified CDT physical therapy protocol, based on Godoy's Method, was applied to all study participants. This protocol comprised of
  1. Cervical Stimuli 15min
  2. MLD based on Godoy
  3. Mechanical lymphatic drainage with RA Godoy® device
  4. Compression therapy with multilayer and multicomponent bandages during the mechanical lymphatic drainage.
  5. Skin care - before and after the bandages- and therapeutic education.
  6. Put on compression garments
  7. Active movement if possible.
  Interventions: Other: modified CDT physical therapy protocol, based on Godoy's Method

INTERVENTIONS:
Other: modified CDT physical therapy protocol, based on Godoy's Method — modified CDT physical therapy protocol

SUMMARY:
The goal of this observational study or clinical trial is to know evaluate the effects of a modified Complete Decongestive Therapy protocol using the Godoy Method in the postoperative period following lipedema surgery.

The main question it aims to answer are:

* if the treatment is effective on pain reduction, edema resorption, mobility improvement in short term and follow-up at 90 days
* if the treatment is effective on preventing complications of these participants after surgery

Participants have been treated in the lasts years and authors recover information of the effects of the treatment.

Researchers will compare sub-groups of participants depending on the number of physical therapy sessions received

DETAILED DESCRIPTION:
Background: Lipedema is an adipose tissue disorder in women, with an abnormal fat deposition in lower limbs and occasionally upper limbs. The patients present pain, bruising, heaviness, and mobility impairment. It affects them physically and psychologically. Purpose: This study aims to evaluate the effects of a modified CDT protocol using the Godoy Method in the postoperative period following lipedema surgery.

Outcomes: pain (VAS), edema resorption, complications, mobility and patient satisfaction.

A descriptive statistical analysis will be performed using means and standard deviation (quantitative outcomes) and percentages (dichotomous and categorical outcomes). An inferential analysis will be carried out using paired and unpaired T-tests as One-way and repeated measures ANOVA to search for differences between quantitative outcomes. Pearson chi-square will also be used to relate dichotomous and categorical variables in a transversal analysis. All missing values will be excluded from the analysis. In all cases, a P<0.05 value and a 95% confidence interval will be determined forstatistical significance. All statistical analysis will be performed using the Stata® version 14.2 package for MS Windows® version 10.

ELIGIBILITY:
Inclusion Criteria:

* female subject who underwent a lipedema surgery
* recommendation of the surgeon to receive physical therapy

Exclusion Criteria:

* unilateral surgery
* lack of data in the clinical history
* only 1-2 physical therapy sessions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: females from undergon a surgical proceeding for lipedema in two private hospitals in Madrid and were treated in a private physical therapy center. After surgery they were recommended to receive CDT by their surgeons. All participants received the same physical therapy treatment. The study was approved by the Clinical Research Committee of Hospital Universitario Principe de Asturias (CEIm 36/2023).
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Pain VAS scale | 2018-2022
  VAS

SECONDARY OUTCOMES:
edema resorption - volume | 2018-2022
  lower limb edema is measured
complications reported - binary outcome | 2018-2022
  seroma, wound infection, chafing or risk of ulcer, pain, fibrosis, genital edema
mobility - scale | 2018-2022
  1- dependent to move/no improvement, 2-somewhat dependent/minor to medium improvement, 3- independent marked improvement
patient satisfaction | 2018-2022
  binary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ester Cerezo Tellez, Alcalá de Henares, Madrid, Spain